CLINICAL TRIAL: NCT06092463
Title: The Intestinal Innate Immune System in Newborns. Development and Inflammation in
Brief Title: The Intestinal Innate Immune System in Newborns. Development and Inflammation in Health and Disease
Acronym: INTINE
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Technical University of Denmark (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lise Aunsholt, senior consultant, Ph.D., Associate Professor, Rigshospitalet, Denmark
Other Study IDs: S-20220057
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Preterm Infants; Term Infants; Necrotising Enterocolitis; Atresia; Bowel; Innate Inflammatory Response
Keywords: IgA; mRNA sequencing; Nutritional support; Bowel habbits
MeSH Terms: conditions — Enterocolitis, Necrotizing; Intestinal Atresia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — faecal material and intestinal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preterm infants: Infants will be included just after birth after obtained consent based on written and verbal information. Fecal samples will be collected from day 1 of life and weekly for the following weeks until discharge to investigate the composition of the fecal microbiome in relation to the development of NEC and the effect of medical therapy.
  In case of development of NEC with the need for surgery the affected intestine will be resected and stomas will be established. Samples of fecal content and tissue is collected from intestine proximal and distal to divided intestine. At time of reversal of stomas, again tissue will be collected both proximal and distal from division to investigate the development of the intestine during early life as well as potential nutritional effects on intestinal maturity. Infants who do not undergo surgery serve as controls, those who are treated for NEC with antibiotics only, will be included in a sub analysis comparing the microbiome of infants who need surgery.
- Newborn and children up to 1 year of age: Infants with congenital malformations will have to undergo scheduled surgery to resect and/or anastomose the affected area of the intestine and some will receive a stoma that needs later reversal. At primary surgery fecal samples and intestinal tissue will be collected proximal and distal to the pathology. In cases with a stoma, and when the child will undergo later reversal surgery, tissue samples from the proximal and distal ends of the intestine will be collected together with fecal samples.

SUMMARY:
The goal of this observational study is to determine the normal development of the human intestinal immune system in premature and mature neonatal life and to determine the pathophysiology behind life-threatening gastrointestinal diseases that appear during early life. The main questions aim to answer are:

* to determine the normal development of the human intestinal immune system in premature and mature neonatal life and to determine the pathophysiology behind life-threatening gastrointestinal diseases that appear during early life.
* is to investigate the development of the immune system in relation to enteral nutrition during the neonatal period.

Participants will be asked to give faecal samples from day 1 of life and weekly for the following weeks until discharge (preterm infants). Further, surgery faecal samples and intestinal tissue will be collected proximal and distal to the pathology. In cases with a stoma, and when the child will undergo later reversal surgery, tissue samples from the proximal and distal ends of the intestine will be collected together with fecal samples (preterm and children up to 1 year of age who need to undergo intestinal surgery due to atresia).

DETAILED DESCRIPTION:
1. NEC Study 1.1. Inclusion criteria Premature infants born < GA week 32. The total number to be included will be 200 1.2. Exclusion criteria Premature born with congenital diseases or other serious conditions may defer participation.

Situations where collection of tissue at surgery is impossible or problematic e.g. due to the remaining length of the vital intestine are evaluated to be too short according to the discretion of the operating surgeon.

1.3. Study design Infants will be included just after birth after obtaining consent based on written and verbal information. Faecal samples will be collected from day 1 of life and weekly for the following weeks until discharge to investigate the composition of the faecal microbiome in relation to the development of NEC and the effect of medical therapy.

In case of the development of NEC with the need for surgery, the affected intestine will be resected, and stomas will be established. Samples of faecal content and tissue are collected from the intestine proximal and distal to the divided intestine. At the time of reversal of stomas, the tissue will be collected both proximal and distal from division to investigate the development of the intestine during early life as well as potential nutritional effects on intestinal maturity. Infants who do not undergo surgery serve as controls, those who are treated for NEC with antibiotics only, will be included in a sub-analysis comparing the microbiome of infants who need surgery.

1.4. Sampling 1.4.1. Fecal samples Faecal samples are collected as soon as possible after birth and once weekly until discharge. Faeces is scraped off the diaper as soon as this appears. The amount must match a fingernail. Two samples are collected at each time point. Faces will be stored in an appropriate tube, after collection, the content is mixed with a buffer (saline) 1:2 before freezing at -600 degrees C. Fecal content collected at primary surgery and at stoma reversal, samples are prepared similarly.

1.4.2. Intestinal samples At surgery a tissue sample from the proximal and distal end of the resected intestine and remnant intestine are taken and snap-frozen immediately after collection and stored at -800 C. To be able to collect as many tissue samples as possible, our strategy will be to snap freeze at least 4 samples (approximately 1 cm2) of the resected tissue; 2 from the healthy site and 2 from the diseased site of the intestine. One or more samples will be prepared for fresh analysis at DTU (only from infants from Rigshospitalet). At stoma reversal tissue will be taken from the stoma site and the proximal end of the diverted intestine. All tissue will be transferred to a biobank hosted by OPEN at Odense University Hospital.

1.5. Outcomes 1.5.1. Primary To investigate the role of microbiota in the development of NEC and associated changes in the intestinal immune system in those who will be operated 1.5.2. Secondary: Demographics such as GA, BW, type of birth and Apgar score Clinical: Growth, type of nutrition, number of days on TPN, number of days with central venous catheter and medical treatment. 1.6. Information and consent Premature infants admitted to either the Department of Intensive Care of Infants and Toddlers, Rigshospitalet or the Department of Neonatology, OUH will be screened for eligibility. The necessary information will be handed over to the researchers. For children that fulfil the inclusion criteria, the parents will be approached and informed about the project and asked for participation in the study and their informed written consent. The parents' consent to participate in the study must be documented in the patient's electronic medical record. Informed consent must be obtained prior to the collection of any samples for the project. If the parents wish, they can have access to a bystander from among the personnel with no direct relation to the research project, and they will also be given the possibility to bring along an assessor. Besides written and oral information about the study the pamphlet "Før du beslutter dig: Om at være forsøgsperson i sundhedsvidenskabelige forsøg" from VEK, together with the pamphlet "Forsøgspersonens rettigheder i et sundhedsvidenskabeligt forskningsprojekt'' will be delivered to the parents. If the parents consent, they will receive a copy of the informed consent form.

If possible, a consideration period of 24 hours will be offered before signing the informed consent, in which case a new meeting (the screening) will be scheduled. If participants do not require time for consideration, the declaration of informed consent may be signed immediately after the information meeting by the participant's mother or the parents of the participant and the investigator (or the research team who have had this responsibility assigned by the investigator). When the informed consent is signed, the participant will be offered a copy. Signed informed consent is a prerequisite for screening or any study-related procedures to start.

1. Atresia study 1.1. Inclusion All newborns and children up to 1 year of age need to undergo intestinal surgery due to atresia at any site of the intestine. An inclusion of a total of 75 patients is anticipated.

1.2. Exclusion For infants and children intestinal tissue sampling would compromise surgery and the health of the patient.

1.3. Study Design Infants with congenital malformations will have to undergo scheduled surgery to resect and/or anastomose the affected area of the intestine, and some will receive a stoma that needs later reversal. At primary surgery, faecal samples and intestinal tissue will be collected proximal and distal to the pathology. In cases with a stoma, and when the child will undergo later reversal surgery, tissue samples from the proximal and distal ends of the intestine will be collected together with faecal samples.

1.4. Sampling 1.4.1. Fecal samples Fecal samples are collected as soon as possible after primary operation and once weekly until discharge. Faeces is scraped of the diaper as soon as this appears. The amount must match a fingernail. Two samples are collected at each time point. Faeces will be stored in an appropriate tube, after collection, the content is mixed with a buffer (saline) 1:2 before freezing at -600 degrees C. Fecal content collected at primary surgery and at stoma reversal, samples are prepared similarly.

1.4.2. Intestinal samples At surgery 2 or more tissue samples from the proximal and distal intestines will be collected. To be able to collect as many tissue samples as possible, our strategy will be to snap freeze at least 4 samples (approximately 1 cm2) of the resected tissue; 2 from the proximal and distal part, respectively. One or more samples will be prepared for fresh analysis at DTU (only from infants at Rigshospitalet). The same procedure will be performed at stoma reversal. All tissue will after termination of the study be transferred to a biobank hosted by OPEN at Odense University Hospital.

1.5. Outcomes: 1.5.1. Primary Constitution and development of the intestinal immune system and intestinal bacterial colonization over time 1.5.2. Secondary Demographics such as GA, BW, type of birth and Apgar score Clinical: Growth, type of nutrition, medical treatment, and disease course. 1.6. Information and consent Infants born with a congenital malformation in the gastrointestinal tract that needs surgery will be screened for eligibility. The necessary information will be handed over to the researchers. For children that fulfil the inclusion criteria, the parents will be approached and informed about the project and asked for participation in the study and their informed written consent. The parents' consent to participate in the study must be documented in the patient's electronic medical record. Informed consent must be obtained prior to the collection of any samples for the project Written and oral information will be carried out by staff from either the Department of IntensiveCare of Infants and Toddlers, Rigshospitalet, Department of Paediatric Surgery, Rigshospitalet, Department of Paediatric Surgery, OUH or the Department of Neonatology, OUH. If the family wishes, they can have access to a bystander from among the staff with no direct relation to the research project, and they will also be given the possibility to bring along an assessor. Besides written and oral information about the study, the pamphlet "Før du beslutter dig: Om at være forsøgsperson i sundhedsvidenskabelige forsøg" from VEK, together with the pamphlet "Forsøgspersonens rettigheder i et sundhedsvidenskabeligt forskningsprojekt'' will be delivered to the parents. If the parents consent, they will receive a copy of the informed consent form.

If possible, a consideration period of some hours during the waiting period for surgery will be offered before signing the informed consent. If participants do not require time for consideration, the declaration of informed consent may be signed immediately after the information meeting by the participant's mother or the parents of the participant and the investigator (or the research team who have had this responsibility assigned by the investigator). When the informed consent is signed, the participant will be offered a copy. Signed informed consent is a prerequisite for any study-related procedures to start.

ELIGIBILITY:
Inclusion Criteria:

NEC study

* Premature infants born < GA week 32 Atresia study
* All newborn and children up to 1 year of age who needs to undergo intestinal surgery due to atresia at any site of the intestine.

Exclusion Criteria:

NEC study - Premature born with congenital diseases or other serious conditions which may defer participation. Situations where collection of tissue at surgery is impossible or problematic e.g. due to remaining length of vital intestine is evaluated to be too short according to the discretion of the operating surgeon.

Atresia study

-Infants and children where intestinal tissue sampling would compromise surgery and the health of the patient subsequent.

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants and children up to 1 year of age
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
If faecal IgA may be an early marker of NEC in preterm infants | 6 years
  IgA measures in repetative faecal samples from admission till disease or GA 34 weeks in no-NEC infants
Development of the intestinal immune system over time | 6 years
  mRNA sequencing of intestinal tissue from preterm infants exposed to surgery due to NEC and compared to intestinal tissue removed from term infants undergoing surgery due to atresia.

SECONDARY OUTCOMES:
Nutritional impact on intestinal development | 6 years
  Comparison of tissue removed at primary surgery in preterm with NEC and at later stomareversal. measurements are:Growth in kg, type of nutrition (MOM, DHM or Formula), number of days on TPN, number of days with central venous catheter and medical treatment.
Bowel habits in preterm infants as marker for later intestinal disease | 6 years
  Comparison of meconium passage (measured in hours), faecal scores (using Amsterdam stool scale) and use of laxative (prescription day, number of days, and type of laxative) in preterm who remain intestinal healthy to those who develop medical and surgical NEC or SIP

CONTACTS AND LOCATIONS:
Overall Officials: Lise Aunsholt, ph.d., Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - University hospital of sounthen denmark, Odense

IPD SHARING:
Plan to Share IPD: No